CLINICAL TRIAL: NCT04023539
Title: Evaluation of the Effect of Cinnamomum Zeylanicum on Glycemic Levels of Mexican Adult Patients With Type 2 Diabetes at 3 Months: Randomized Clinical Trial
Brief Title: Effect of Cinnamomum Zeylanicum on Glycemic Levels of Adult Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Julio Alfredo Garcia Puga, Principal Investigator, Universidad de Sonora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cinnamon-T2D-MEX-2019
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes
Keywords: Cinnamon; Type 2 diabetes; Diabetes; México; Cinnamomum zeylanicum; Randomized Controlled Trial; Glycated hemoglobin; Glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial This is a simple blind randomized clinical trial with patients with type 2 diabetes, the subjects will be divided into two groups, the intervention supplemented with 2 g daily of cinnamomum zeylanicum orally (capsules) and the control group with a placebo. There will be a follow-up of 3 months every two weeks to measure the variables of interest in the study.
Who Masked: Participant
Masking Description: A simple blinding (participants blinded to the belonging group). The person who will randomize the participants will not be involved in the recruitment of participants. This will be done when we have the total sample of participants.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Daily supplement of 2 g cinnamomum zeylanicum orally (capsules) for a period of 90 days
  Interventions: Dietary Supplement: Cinnamomum zeylanicum
- Control group (Placebo Comparator): Daily placebo capsules orally (wheat flour without any active compound) for a period of 90 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Cinnamomum zeylanicum — Capsules of 2 g cinnamomum zeylanicum orally
  Arms: Intervention group
Other: Placebo — Placebo capsules
  Arms: Control group

SUMMARY:
Type 2 Diabetes (T2D) is protected against chronic hyperglycemia. This is one of the main causes of death in the country, being a public health problem worldwide. Some studies have shown that herbal products have beneficial effects in patients with diabetes by improving the metabolism of glucose and lipids. Cinnamomum Zeylanicum (C.Z.), colloquially cinnamon, is one of the components of the diet that has active biological substances with insulin mimetic properties. In Mexico, little has been investigated about the use of this therapy. Previous studies do not conclude if there is a statistically significant effect in the glycemic control of patients with diabetes. Therefore, it is proposed to evaluate the effect of the supplement consumption of C.Z. 3 months compared to a control group on the change in glycated hemoglobin (HbA1c) in Mexican adults with T2D. This is a randomized, single-blind clinical trial with T2D patients from the clinic CAAPS . Those that are divided into: intervention group with supplement of 2g daily C.Z. Oral route (capsules) for 90 days, and control group with placebo. The figures will be recorded: HbA1c, fasting plasma glucose, blood pressure, cholesterol, HDL, LDL, triglycerides, waist circumference, weight and body mass index.

DETAILED DESCRIPTION:
Cinnamon, in in vitro and in vivo studies, has been shown to have biologically active substances with mimetic properties of insulin. In 1990 an unidentified component of cinnamon was extracted and named as an insulin-enhancing factor. The components of cinnamon bark oil (Ceylon) contain cinnamaldehyde (75%), cinnamyl acetate (5%), caryophyllene (3.3%), linalool (2.4%) and eugenol (2.2%). It is believed that the modality in which cinnamon expresses its effect on blood glucose can be attributed to its active component cinnamaldehyde.

Within the 250 species of the Cinnamomum genus there are four types that are used as spice, the Cinnamomum Zeylanicum or Sri Lanka (also known as C. verum Ceylon) commonly referred to as "true cinnamon"; three very popular spices related to C. cassia are C. aromaticum (cinnamon china), C. loureirii (cinnamon vietnamese) and C. burmanni (cinnamon indonesia).

One important difference between "true cinnamon" and cinnamon cassia is its coumarin content. The content of coumarin in cinnamomum zeylanicum is too low to cause health risks, while the level of coumarin in Cinnamomum aromaticum appears to be much higher and may pose health risks if consumed in larger quantities and on a regular basis. The use of cinnamon cassia as a regular supplement with meals is not recommended or the daily dose has been restricted in many countries due to the toxic effects of Cinnamomum aromaticum on the liver and coagulation. In contrast, cinnamomum zeylanicum has been shown to contain a lower amount of coumarin, and therefore it may be possible to use it at higher doses without toxic effects for longer periods. In vivo studies with cinnamomum zeylanicum have not shown significant adverse effects or toxicity in liver, kidney and / or pancreas.

In a systematic review it was concluded that the evidence available in vitro and in vivo suggests that cinnamomum zeylanicum has antimicrobial, antiparasitic, anti-inflammatory and antioxidant properties. The authors also indicated that cinnamomum zeylanicum appears to lower blood glucose, serum cholesterol, and blood pressure, suggesting beneficial cardiovascular effects.

The mechanism of this hypoglycaemic action is not entirely clear, but can be attributed to an increase in serum insulin levels, storage of liver glycogen, better signaling of the insulin receptor, an insulinomimetic effect, or reduction of alpha activity intestinal -glucosidase. In clinical terms, these actions could lead to improvements in glycemic control and insulin sensitivity, and a possible reduction in the complications of diabetes.

In Mexico, little has been investigated on the use of this alternative therapy. In other countries, such as the United States, the United Kingdom, China, Pakistan and Germany, studies have been conducted on the potential effects of cinnamomum in in vitro, in vivo and in human studies. The effect of C. zeylanicum on glycemic control is inconclusive due to the contradictory results of the literature, some authors found statistically significant changes in glycosylated hemoglobin or fasting plasma glucose in randomized clinical trials compared with a placebo group. On the other hand, several authors report not having found significant changes in glucose levels in the study subjects.

In the case of the Mexican population, no scientific studies were found that address the use of cinnamomum as an alternative therapy-alone or combined-in the control of glycemic levels in patients with diabetes. Therefore, in this study we propose to evaluate the effect of cinnamomum zeylanicum supplement consumption at 3 months compared to a control group (placebo) on the change in HbA1c in Mexican adults with T2D.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a prior medical diagnosis of T2D
* Mexican adults (> 18 years)
* Treatments only with oral hypoglycemic agents
* HbA1c >6.5% and <10%
* Attendees to two participating primary health care centers.

Exclusion Criteria:

* Patients who have an allergy to cinnamon or wheat flour.
* Treatments with insulin
* Gastrointestinal problems or any condition in cinnamon is not well tolerated or contraindicated
* Cardiovascular, hepatic or renal disease.
* Use of addictive substances as drugs.
* Pregnant or lactation
* Psychiatric condition that prevents adherence to treatment
* Use of a supplement with an effect on glucose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | baseline to 3 months
  Change in glycated hemoglobin

SECONDARY OUTCOMES:
Fasting plasma glucose | baseline to 3 months
  Change in fasting plasma glucose
Total cholesterol | baseline to 3 months
  Change in total cholesterol
HDL | baseline to 3 months
  Change in HDL Cholesterol
LDL | baseline to 3 months
  Change in LDL Cholesterol
Triglycerides | baseline to 3 months
  Change in Triglycerides
Weight | baseline to 3 months
  Change in Weight
Waist circumference | baseline to 3 months
  Change in waist circumference
Body Mass Index | baseline to 3 months
  Change in the Body Mass Index
Blood pressure | baseline to 3 months
  Change in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Julio Alfredo García Puga, Ph.D., Principal Investigator — Universidad de Sonora
Locations (2):
- Mexico (2):
  - C.A.A.P.S., Hermosillo, Sonora
  - ISSSTE Family Medicine Clinic, Hermosillo, Sonora

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranasinghe P, Perera S, Gunatilake M, Abeywardene E, Gunapala N, Premakumara S, Perera K, Lokuhetty D, Katulanda P. Effects of Cinnamomum zeylanicum (Ceylon cinnamon) on blood glucose and lipids in a diabetic and healthy rat model. Pharmacognosy Res. 2012 Apr;4(2):73-9. doi: 10.4103/0974-8490.94719. PMID 22518078
- [Background] Sangal A. Role of cinnamon as beneficial antidiabetic food adjunct: A review. Advaces in Applied Science Research. 2010;2(4):440-50
- [Background] Allen RW, Schwartzman E, Baker WL, Coleman CI, Phung OJ. Cinnamon use in type 2 diabetes: an updated systematic review and meta-analysis. Ann Fam Med. 2013 Sep-Oct;11(5):452-9. doi: 10.1370/afm.1517. PMID 24019277
- [Background] Costello RB, Dwyer JT, Saldanha L, Bailey RL, Merkel J, Wambogo E. Do Cinnamon Supplements Have a Role in Glycemic Control in Type 2 Diabetes? A Narrative Review. J Acad Nutr Diet. 2016 Nov;116(11):1794-1802. doi: 10.1016/j.jand.2016.07.015. Epub 2016 Sep 8. PMID 27618575
- [Background] Lungarini S, Aureli F, Coni E. Coumarin and cinnamaldehyde in cinnamon marketed in Italy: a natural chemical hazard? Food Addit Contam Part A Chem Anal Control Expo Risk Assess. 2008 Nov;25(11):1297-305. doi: 10.1080/02652030802105274. PMID 19680836
- [Background] Ranasinghe P, Jayawardena R, Pigera S, Wathurapatha WS, Weeratunga HD, Premakumara GAS, Katulanda P, Constantine GR, Galappaththy P. Evaluation of pharmacodynamic properties and safety of Cinnamomum zeylanicum (Ceylon cinnamon) in healthy adults: a phase I clinical trial. BMC Complement Altern Med. 2017 Dec 28;17(1):550. doi: 10.1186/s12906-017-2067-7. PMID 29282046
- [Background] Ranasinghe P, Pigera S, Premakumara GA, Galappaththy P, Constantine GR, Katulanda P. Medicinal properties of 'true' cinnamon (Cinnamomum zeylanicum): a systematic review. BMC Complement Altern Med. 2013 Oct 22;13:275. doi: 10.1186/1472-6882-13-275. PMID 24148965
- [Background] Leach MJ, Kumar S. Cinnamon for diabetes mellitus. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007170. doi: 10.1002/14651858.CD007170.pub2. PMID 22972104
- [Background] Akilen R, Tsiami A, Devendra D, Robinson N. Glycated haemoglobin and blood pressure-lowering effect of cinnamon in multi-ethnic Type 2 diabetic patients in the UK: a randomized, placebo-controlled, double-blind clinical trial. Diabet Med. 2010 Oct;27(10):1159-67. doi: 10.1111/j.1464-5491.2010.03079.x. PMID 20854384
- [Background] Khan A, Safdar M, Ali Khan MM, Khattak KN, Anderson RA. Cinnamon improves glucose and lipids of people with type 2 diabetes. Diabetes Care. 2003 Dec;26(12):3215-8. doi: 10.2337/diacare.26.12.3215. PMID 14633804
- [Background] Khan R, Khan Z, Hussain Shah S. Cinnamon May Reduce Glucose, Lipid and Cholesterol Level in Type 2 Diabetic Individuals. Pakistan J Nutr. 2010;9(5):430-3
- [Background] Lu T, Sheng H, Wu J, Cheng Y, Zhu J, Chen Y. Cinnamon extract improves fasting blood glucose and glycosylated hemoglobin level in Chinese patients with type 2 diabetes. Nutr Res. 2012 Jun;32(6):408-12. doi: 10.1016/j.nutres.2012.05.003. Epub 2012 Jun 14. PMID 22749176
- [Background] Sharma P, Sharma S, Agrawal RP, Agrawal V, Singhal S. A randomised double blind placebo control trial of cinnamon supplementation on glycemic control and lipid profile in type 2 diabetes mellitus. Aust J Herbal Med. 2012;24(1):52-7.
- [Background] Mang B, Wolters M, Schmitt B, Kelb K, Lichtinghagen R, Stichtenoth DO, Hahn A. Effects of a cinnamon extract on plasma glucose, HbA, and serum lipids in diabetes mellitus type 2. Eur J Clin Invest. 2006 May;36(5):340-4. doi: 10.1111/j.1365-2362.2006.01629.x. PMID 16634838
- [Background] Crawford P. Effectiveness of cinnamon for lowering hemoglobin A1C in patients with type 2 diabetes: a randomized, controlled trial. J Am Board Fam Med. 2009 Sep-Oct;22(5):507-12. doi: 10.3122/jabfm.2009.05.080093. PMID 19734396
- [Background] Blevins SM, Leyva MJ, Brown J, Wright J, Scofield RH, Aston CE. Effect of cinnamon on glucose and lipid levels in non insulin-dependent type 2 diabetes. Diabetes Care. 2007 Sep;30(9):2236-7. doi: 10.2337/dc07-0098. Epub 2007 Jun 11. No abstract available. PMID 17563345
- [Background] Mirfeizi M, Mehdizadeh Tourzani Z, Mirfeizi SZ, Asghari Jafarabadi M, Rezvani HR, Afzali M. Controlling type 2 diabetes mellitus with herbal medicines: A triple-blind randomized clinical trial of efficacy and safety. J Diabetes. 2016 Sep;8(5):647-56. doi: 10.1111/1753-0407.12342. Epub 2015 Dec 1. PMID 26362826
- [Background] Suppapitiporn S, Kanpaksi N, Suppapitiporn S. The effect of cinnamon cassia powder in type 2 diabetes mellitus. J Med Assoc Thai. 2006 Sep;89 Suppl 3:S200-5. PMID 17718288
- [Background] Vafa M, Mohammadi F, Shidfar F, Sormaghi MS, Heidari I, Golestan B, Amiri F. Effects of cinnamon consumption on glycemic status, lipid profile and body composition in type 2 diabetic patients. Int J Prev Med. 2012 Aug;3(8):531-6. PMID 22973482
- [Background] Vanschoonbeek K, Thomassen BJ, Senden JM, Wodzig WK, van Loon LJ. Cinnamon supplementation does not improve glycemic control in postmenopausal type 2 diabetes patients. J Nutr. 2006 Apr;136(4):977-80. doi: 10.1093/jn/136.4.977. PMID 16549460